CLINICAL TRIAL: NCT04433741
Title: Apply the Pharmacodynamic Model of Peripheral Oxytocin Action to a Multimodal Stimulus That Increases (Heat) or Decreases (Vibration) Pain Perception
Brief Title: Apply the PD Model of Peripheral Oxytocin Action to a Multimodal Stimulus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was never initiated and has been withdrawn and replaced with a new protocol.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00066443
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Cross over model: each participant will be randomized to receive oxytocin and placebo in a random order
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, outcomes assessor and investigator will be blinded to the randomization order. Research pharmacist will prepare each infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oxytocin First, then Placebo (Other): Oxytocin administered intravenously for the first half of the study and then will receive intravenous placebo for the second half.
  Interventions: Drug: Oxytocin; Drug: Placebo
- Placebo, Then Oxytocin (Other): Placebo administered intravenously for the first half of the study and then will receive intravenous oxytocin for the second half.
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Oxytocin administered intravenously
  Other Names: Pitocin
Drug: Placebo — Placebo administered intravenously

SUMMARY:
This is a study of participants that will receive an intravenous (IV) infusion of oxytocin (naturally occurring hormone that is made in the brain).

In this study healthy volunteers are recruited. Each study participant will have an IV catheter placed. After placement of the IV catheter oxytocin will be given by IV infusion of oxytocin or placebo (inactive solution). The investigators will perform some tests to evaluate how oxytocin changes perceptions on the skin. The investigators will study a painful perception by placing a probe on the skin and heating it to 116.6 degrees Fahrenheit for 30 seconds and a vibratory stimulus will be applied to the forearm with vibration begun at a 1 kHz frequency and decreased at a rate of 25 Hz/sec until the subject first perceives the vibration. Each study participant will score any pain that is experienced on a 0 to 10 scale and will report when the vibration is detected. Each participant will receive oxytocin and placebo in a random order and will be blinded to group they are receiving.

DETAILED DESCRIPTION:
The investigators aim to create pharmacokinetic/pharmacodynamic (PK/PD) models for oxytocin action at peripheral sites and at central sites as they relate to sensory transmission and pain. This is the last of 4 studies to accomplish generation, validation, and application of a PK/PD model for oxytocin in the periphery. Its goal is to apply the PK/PD model generated in previous protocols and Validate a pharmacodynamic model of oxytocin for peripheral analgesic effects to a more complex sensory stimulus that stimulates nerve fibers which result in pain from a heat stimulus and those which reduce pain from vibration, similar to brushing or rubbing an area of pain. The investigators do this because oxytocin in animals affects these nerve fibers in the periphery in different ways - it increases the activity of the vibration/rubbing sensitive fibers and decreases the activity of the pain fibers. As such, The investigators expect that the effect of oxytocin on pain from this mixed stimulus of heat and vibration will be much more pronounced than that seen with the purely painful stimulus used in previous studies in this series.

This is a double-blind, crossover study in which oxytocin or placebo is infused. In this study healthy people are recruited for a 2 day double-blind, crossover study. They will come to the Clinical Research Unit and one intravenous catheter (IV) inserted in the forearm for oxytocin or placebo infusion. Participants will be given a steady rate intravenous infusion of oxytocin at a targeted dose or placebo for 30 minutes. At 5, 15, and 30 minutes after starting the infusion, pain report to the 47°Celsius, 30-second stimulus alone or with ½ VT vibration (randomized order) will be obtained. Participants will return at least 24 hours later and receive the opposite infusion and testing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 and < 75 years of age, Body Mass Index (BMI) <40.
2. Generally in good health as determined by the Principal Investigator based on prior medical history, American Society of Anesthesiologists physical status 1 or 2.
3. For healthy volunteers, normal blood pressure (systolic 90-140 mmHg; diastolic 50-90 mmHg) resting heart rate 45-100 beats per minute) without medication.
4. Female subjects of child-bearing potential and those < 1 year post-menopausal, must be practicing highly effective methods of birth control such as hormonal methods (e.g., combined oral, implantable, injectable, or transdermal contraceptives), double barrier methods (e.g., condoms, sponge, diaphragm, or vaginal ring plus spermicidal jellies or cream), or total abstinence from heterosexual intercourse for a minimum of 1 full cycle before study drug administration.

Exclusion Criteria:

1. Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
2. Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
3. Women who are pregnant (positive result for serum pregnancy test at screening visit), women who are currently nursing or lactating, women that have been pregnant within 2 years
4. Subjects with neuropathy, chronic pain, diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Heat pain with vibration | Baseline before infusion
  Pain at the end of 30 sec of heating the skin to 47 degrees C with simultaneous vibration will be determined. Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Heat pain with vibration | 5 minutes post infusion initiation
  Pain at the end of 30 sec of heating the skin to 47 degrees C with simultaneous vibration will be determined. Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Heat pain with vibration | 15 minutes post infusion initiation
  Pain at the end of 30 sec of heating the skin to 47 degrees C with simultaneous vibration will be determined. Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Heat pain with vibration | 30 minutes post infusion initiation
  Pain at the end of 30 sec of heating the skin to 47 degrees C with simultaneous vibration will be determined. Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.

SECONDARY OUTCOMES:
Heat pain without vibration | Baseline
  Pain at the end of 30 sec of heating the skin to 47 degrees C will be determined. Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Heat pain without vibration | 5 minutes post infusion initiation
  Pain at the end of 30 sec of heating the skin to 47 degrees C will be determined. Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Heat pain without vibration | 15 minutes post infusion initiation
  Pain at the end of 30 sec of heating the skin to 47 degrees C will be determined. Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Heat pain without vibration | 30 minutes post infusion initiation
  Pain at the end of 30 sec of heating the skin to 47 degrees C will be determined. Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No